CLINICAL TRIAL: NCT04644289
Title: Window-of-opportunity Proof-of-concept, Non-randomized, Open-label Phase II Trial of Olaparib Given Alone (Cohort A) or in Combination With Durvalumab (Cohort B) Prior to Primary Debulking Surgery in Histologically Proven High-grade Epithelial Ovarian Cancer (EOC)
Brief Title: WoO: Window of Opportunity Trial of Olaparib and Durvalumab in Histologically Proven EOC
Acronym: WoO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 27; 2020-005101-12 (EudraCT Number); 2024-511780-28-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-11; First posted 2020-11-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer; Olaparib; Durvalumab
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — olaparib; durvalumab

STUDY DESIGN:
Intervention Model Description: Patients will be treated in two consecutive cohorts (A, B) of 15 to 30 (cohort A) and 30 (cohort B) patients each, with A) olaparib alone or B) olaparib in combination with durvalumab. Treatment allocation will take please in two consecutive cohorts rather than by randomization. This will allow to evaluate the safety and feasibility in a step-wise approach. A trial steering committee (TSC) meeting will take place between the cohorts to review safety and feasibility prior to starting the second cohort. The safety follow-up of the first cohort will take 90 days as of the first dose of therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cohort A - olaparib monotherapy (Other): Olaparib tablets 2 × 300mg per day for 3 weeks (max. 28 days) prior to surgery until one day prior to surgery or withdrawal of informed consent.
  Patients will receive the indicated standard of care (SoC) chemotherapy plus or minus Bevacizumab as per investigators discretion, followed by SoC maintenance treatment according to the national S3-guideline and treating physician's choice.
  They can be offered:
  For patients in cohort A who have received all possible licensed treatment regimens according to the national guideline or for whom further licensed treatment options are not available or contraindicated, Olaparib may be offered as investigational maintenance therapy for up to 24 months.
  Interventions: Drug: olaparib
- cohort B - olaparib + durvalumab combination (Other): Olaparib tablets 2 × 300mg per day for 3 weeks (max. 28 days) plus Durvalumab 1500mg iv as a single dose prior to surgery (corresponding to 1 single cycle).
  Patients will receive the indicated standard of care (SoC) chemotherapy plus or minus Bevacizumab as per investigators discretion, followed by SoC maintenance treatment according to the national S3-guideline and treating physician's choice.
  They can be offered:
  Patients in cohort B may be offered Durvalumab 1120mg iv Q3W during chemotherapy treatment phase in combination with bevacizumab (unless contraindicated) and as maintenance for a total of up to 24 months (1120mg Q3W) in combination with Bevacizumab (for a total of 15 months, unless contraindicated) and Olaparib for a total of 24 months. For HRD-positive patients Durvalumab will be an investigational agent; for HRD-negative patients Durvalumab and Olaparib will be investigational agents.
  Interventions: Drug: olaparib; Drug: durvalumab

INTERVENTIONS:
Drug: olaparib — Olaparib tablets are administrated orally 300 mg twice daily.
  Other Names: Lynparza
Drug: durvalumab — Durvalumab is administered 1500mg iv as a single dose prior to surgery (corresponding to 1 single cycle) .
  Other Names: Imfinzi
  Arms: cohort B - olaparib + durvalumab combination

SUMMARY:
This is a multi-center, prospective, open-label, phase II trial. Patients with suspected advanced ovarian cancer planned to undergo diagnostic laparoscopy for histologic confirmation and evaluation of disease spread will be registered into the trial after providing a 1st written informed consent.

DETAILED DESCRIPTION:
In total, 60 patients are planned to be enrolled in 2 consecutive cohorts (30 patients per cohort) into the trial.

After histologic confirmation of high-grade epithelial non-mucinous, non-clear cell ovarian cancer, patients will be treated in two consecutive cohorts (A, B) of 30 patients each, with

A) olaparib alone or B) olaparib in combination with durvalumab

Treatment allocation will take place in two consecutive cohorts rather than by randomization. This will allow to evaluate the safety and feasibility in a stepwise approach. A trial steering committee (TSC) meeting will take place between the cohorts to review safety and feasibility prior to starting the second cohort. The safety follow-up of the first cohort will take 90 days as of the first dose of therapy.

Post chemo maintenance:

After completion of first-line chemotherapy patients who have not progressed during first-line chemotherapy will receive the indicated standard maintenance treatment according to the national S3-guideline and treating physician's choice. For patients who have received all possible licensed treatment regimens according to the national guideline or for whom further licensed treatment options are unavailable or contraindicated, Olaparib may be offered as investigational maintenance therapy for up to 24 months. In cohort B, patients will be offered Durvalumab as an investigational therapy in combination with Standard of Care (SoC) chemotherapy and Bevacizumab, followed by a Durvalumab maintenance therapy for a total of 24 months as an investigational therapy in combination with SoC Bevacizumab and Olaparib. Patients for whom the choice of maintenance therapy is Niraparib or who don´t receive Bevacizumab cannot receive Durvalumab maintenance in combination unless they have a contraindication to Bevacizumab, in which case Durvalumab can be offered in combination with SoC chemotherapy and as maintenance therapy in combination with Olaparib. In HRD-negative patients who are selected to receive Bevacizumab maintenance, both Olaparib and Durvalumab will be investigational agents. In HRD-positive patients who are selected to receive Bevacizumab and Olaparib, only Durvalumab will be an investigational agent. The data supporting the rationale and also safety of the combination of Durvalumab, Bevacizumab and Olaparib are based on the randomized, placebo-controlled phase III AGO-OVAR 23/DUO-O study.

ELIGIBILITY:
Inclusion Criteria:

WoO pre-treatment (screening phase):

1. Patients with presumed and previously untreated advanced stage ovarian cancer planned to undergo laparoscopy for histologic diagnosis and treatment planning
2. Patients willing and able to comply with the study protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
3. Patients able and willing to provide fresh frozen biopsy samples from laparoscopy as well as primary debulking for translational endpoints as well as serial liquid biopsies
4. Patients able and willing to provide formaldehyde-fixed paraffin embedded (FFPE) tissue samples from laparoscopy and primary debulking surgery
5. Patients aged ≥18 years
6. Patients must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
7. Provision of signed and dated, written ICF for the mandatory biomarker and genetic re-search as well as the clinical/therapeutic part of the study prior to any mandatory study specific procedures, sampling, and analyses
8. Eastern cooperative oncology group (ECOG) performance status 0-1 (see Appendix 1)
9. Patients must have a life expectancy ≥16 weeks
10. Ability to take oral medication
11. Postmenopausal or evidence of non-childbearing status for women of childbearing potential (WOCBP): negative serum pregnancy test within 28 days of study treatment and confirmed neagtive urine or serum pregnancy test prior to treatment on day 1.

    Postmenopausal is defined as:
    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
    * radiation-induced oophorectomy with last menses >1 year ago
    * chemotherapy-induced menopause with >1 year interval since last menses
    * surgical sterilisation (bilateral oophorectomy or hysterectomy)
12. Women of childbearing potential (WOCBP) and their partners, who are sexually active, must agree to the use of 2 highly effective forms of contraception in combination. This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 6 months after last dose of study drug(s), or they must totally/truly abstain from any form of sexual intercourse.

    WoO treatment phase:
13. Confirmed advanced (FIGO IIB/III/IV) high-grade, non-mucinous, non-clear cell epithelial ovarian, fallopian tube or primary peritoneal cancer or known (BReast CAncer) BRCA mutation and any histologic type
14. Planned primary debulking surgery after confirmation of diagnosis and disease evaluation during laparoscopy
15. Body weight >30kg
16. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥10.0 g/dL with no blood transfusion in the past 28 days
    * Absolute neutrophil count (ANC) ≥1.5×10^9/L
    * Platelet count ≥100×10^9/L
    * Total bilirubin ≤1.5 × institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST), serum glutamic oxaloacetic transaminase (SGOT) / alanine aminotransferase (ALT), serum glutamic pyruvate transaminase (SGPT) ≤2.5 × institutional upper limit of normal unless liver metastases are present in which case they must be ≤5×ULN. (cave: patients with intrahepatic metastases affecting liver function test might not be candidates for primary debulking surgery)
    * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test:

Estimated creatinine clearance=((140-age [years])*weight (kg))/(serum creatinine (mg/dL)*72)(* 0,85) 17. Patients must have successfully contributed blood and tissue samples as per requirements.

Exclusion Criteria:

Medical conditions:

1. Disease requiring urgent surgical intervention
2. Evidence of significant uncontrolled concomitant disease that could affect compliance with the study protocol
3. Significant uncontrolled symptom burden (e.g. but not necessarily limited to large volume ascites, shortness of breath on exertion, pain requiring opioid medication, signs of (sub)ileus
4. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, recent (within 3 months) myocardial infarction, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
5. Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), stage 1, grade 1 endometrial carcinoma. Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease (optional criteria that is dependent on the patient population under investigation).
6. Resting electrocardiography (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, conges-tive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   a. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with olaparib, durvalumab or the combination may be included only after consultation with the coordinating investigator.
8. Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML).
9. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
10. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
11. Evidence of central nervous system (CNS) or leptomeningeal metastases.
12. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders or any status that might interfere with resorption of the respective study drugs, e.g. parenteral nutrition, short bowel syndrome likely to interfere with absorption of the study medication.
14. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
15. History of active primary immunodeficiency
16. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B or hepatitis C.

    1. Active HBV is defined by a known positive HBsAg result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
    2. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA
17. ECOG performance status (PS) ≥2 or general condition that might interfere with the compliance with the study protocol
18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

    Prior / concomitant therapy:
19. Prior antineoplastic therapy for ovarian, fallopian tube or primary peritoneal cancer
20. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
21. Any concurrent chemotherapy, investigational medicinal product (IMP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
22. Patients planned for neoadjuvant chemotherapy or deemed unresectable at laparoscopy
23. Concomitant use of known strong cytochrome P450 3A (CYP3A) inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
24. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
25. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
26. History of allogenic organ transplantation
27. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
28. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
29. Prior treatment with olaparib or any other poly [ADP-ribose] polymerase (PARP) inhibitor
30. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no. 16)

    Other exclusions:
31. Patients who are pregnant or breast-feeding or patients of reproductive potential who are not willing to employ effective birth control from screening to 6 months after the last dose of study drug(s).
32. Involvement in the planning and/or conduct of the study
33. Participation in another interventional clinical study with an investigational product during the last with the last 3 months.
34. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
35. Previous enrolment in the present study.
36. Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

    Additional Durvalumab-specific exclusion criteria for cohort B:
37. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤28 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or pharmacokinetic (PK) properties of an agent, a longer wash-out period will be required.
38. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the coordinating investigator.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the coordinating investigator.
39. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
40. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note: local surgery of isolated lesions for palliative intent is acceptable.
41. History of allogenic organ transplantation.
42. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or wegener syndrome [granulomatosis with polyangiitis, graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
43. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring (Adverse Events) AEs or compromise the ability of the patient to give written informed consent.
44. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IMP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
45. History of leptomeningeal carcinomatosis
46. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
47. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
48. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive hepatitis B virus (HBV) surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-hepatitis-B-core (HBc)] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
49. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
50. Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP. Note: patients, if enrolled, should not receive live vaccine whilst receiving IMP and up to 30 days after the last dose of IMP.
51. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment or other immunotherapies
52. Patients who have received prior anti-programmed cell death-protein 1(PD-1), anti PD-L1 or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4):

    1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    3. Must not have experienced a ≥grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. Note: Patients with endocrine AE of ≤grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if rechallenged, and not currently require maintenance doses of >10 mg prednisone or equivalent per day.
53. Patients planned for neoadjuvant chemotherapy (e.g. but not exclusively due to extend of disease spread or poor general condition etc.).
54. (sub)ileus or signs of malignant bowel obstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the WoO procedure for olaparib alone (cohort a) & olaparib in combination with durvalumab (cohort b) | Between registration into the trial until 60 days after surgery or 60 days after the originally planned surgery date in case of switch of therapeutic strategy.
  Defined as the successful completion of the WoO therapy:
  * Relative dose intensity (RDI) of ≥80%
  * No treatment-related surgical delays
  * Adherence to therapeutic strategy
  * Lack of clinical progression prior to primary debulking surgery
  * No treatment-related toxicities of any grade that in the judgment of the investigator or surgeon significantly interfered with the subject's optimal perioperative management

SECONDARY OUTCOMES:
Safety of the WoO procedure | Between registration into the trial until 60 days after surgery or 60 days after the originally planned surgery date in case of switch of therapeutic strategy.
  Evaluated by the proportion of patients who experience any adverse event (CTCAE v5.0), of a grade ≥3.
Proportion of circulating tumor DNA (ctDNA) Mutation positive patients | At baseline
  Proportion of ctDNA mutation positive patients at baseline above a predefined a cut-off (copies/ml).
CDR21 | At day 21
  Circulating DNA ratio at day 21 (CDR21) defined as the ratio of mutation abundance at day 21 relative to baseline of the mutant ctDNA allele with the highest abundance (mutant copies/ml) at baseline.

OTHER OUTCOMES:
Progression free survival (PFS) | From registration until progression or death or date of LPLV whichever occurs first. Depending on the time point of inclusion into the trial the expected maximum follow-up time for an individual patient might range between 2.5 and 4,6 years.
  Defined as the time from registration into the trial (PIC2) until radiologic progression or progression according to GCIG criteria during routine follow-up or or death without progression or clinical deterioration of performance status with associated signs of disease (e.g. bowel obstruction and non-measurable disease).
PD-L1 expression | At day 21
  Comparing PD-L1 expression between ctDNA responders and non-responders (CDR21 median)

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Marmé, MD, Principal Investigator — Universitätsklinikum Mannheim, Frauenklinik
Locations (6):
- Germany (6):
  - Universitätsklinikum Mannheim GmbH, Frauenklinik, Mannheim, Baden-Wurttemberg
  - Klinikum rechts der Isar, Technische Universität München, Klinik und Poliklinik für Frauenheilkunde, München, Bavaria
  - Mammazentrum HH am Krankenhaus Jerusalem, Gynäkologisches Operationszentrum Hamburg, Hamburg, Hamburg
  - KEM Essen | Evang. Kliniken Essen Mitte, Essen, North Rine-Westphalia
  - Universitätsklinikum Carl Gustav Carus Dresden an der technischen Universität Dresden, Gynäkologisches Krebszentrum und Regionales Brustzentrum Dresden am Universitäts-KrebsCentrum, Dresden, Saxony
  - Charité Berlin, Klinik für Gynäkologie mit Zentrum für onkologische Chirurgie, Berlin, State of Berlin

REFERENCES:
- See also: Homepage of AGO Study Group — http://www.ago-ovar.de/